CLINICAL TRIAL: NCT04431102
Title: The Effects of the Pilates Method on Pelvic Floor Injuries During Pregnancy and Childbirth: A Quasi-experimental Study
Brief Title: Pilates and the Pelvic Floor: A Quasi-experimental Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Huelva (Other)
Responsible Party: Principal Investigator, Mª Carmen Feria Ramírez, Principal investigator, University of Huelva
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CFMP14
Record Dates: First submitted 2020-06-10; First posted 2020-06-16 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Pregnancy; Perineum; Injury; Pilates Method; Episiotomy Wound
Keywords: Nursing; Midwifery; Nurse; Pilates Method; Pelvic floor; Injuries; Episiotomy; Pregnancy
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: The professionals who assessed the progress of labor in the delivery room and completed the medical history did not know whether the woman belonged to the intervention or the control group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PILATES METHOD (Experimental): It was intended the Pilates program were low supervision and easily realizable by all patients, which implied flexibility in the schedule. In this sense the sessions of Pilates was adjusted to these assumptions and the Pilates monitor offered several schedules on diferent days of the week.
  The pregnant women assigned to the intervention group were supervised by the midwifery of reference and trained by a Pilates monitor who explained the training program. The women received eight sessions of Pilates, given with a frequency of two classes per week and one hour of duration during a period of four weeks. The exercises for each session were determined beforehand. In addition, the participants maintained the usual monitoring of pregnancy valued by the reference average, attending the sessions of the maternal education program of their health center.
  The therapeutic control were carried out by telephone call and clinical history review between the eighth and tenth day postpartum.
  Interventions: Other: PILATES METHOD
- MATERNAL EDUCATION (No Intervention): The control group maintained the usual monitoring of pregnancy valued by the reference average, attending the sessions of the maternal education program of their health center.
  Therapeutic control was carried out by phone call and review of the clinical history between the eighth and tenth day postpartum.

INTERVENTIONS:
Other: PILATES METHOD — It is intended that the Pilates program have a duration of four weeks and its realization does not suppose an excessive consumption of resources. Therefore, it must have a series of characteristics: low supervision and easily realizable by all patients, which implies flexibility in the schedule. In this sense the sessions of Pilates is adjusted to these assumptions and the Pilates monitor offers several schedules on diferent days of week.
  The pregnant women assigned to the intervention group will be supervised by the midwifery of reference and trained by a Pilates monitor who will explain the training program and resolve the doubts raised by the women.
  The therapeutic control will be carried out by telephone call and clinical history review between the eighth and tenth day.
  Arms: PILATES METHOD

SUMMARY:
In this paper, it is postulates that in pregnant women, the practice of PM led by a qualified professional for a period of four weeks can reduce the incidence of pelvic floor dysfunction (PFD) by decreasing the number of birth injuries.

DETAILED DESCRIPTION:
It is postulated that in pregnang women, the practice of PM can reduce the severity of birth injuries.

Our main objective was to determine the effectiveness of a PM program to reduce the incidence and degree of intrapartum perineal injuries as a way to reduce the incidence of female PFD.

Secondary objectives were:

Assess the role of a MP program on the systolic and diastolic blood pressure. Determine the effect of a MP program on body weight (BMI).

It is a parallel group clinical trial with an allocation ratio of 1:2.

All pregnant women will be informed about the nature of the clinical trial. There will be no differences in the pregnant´s follow-up because it will be performed by two same Pilates monitor with the same formation.

Once the pregnant women is assigned to an arm of the study, those assigned to the intervention group will be sent to the Pilates monitor to explain and initiate the exercise of MP program while the control group will be informed to maintain their usual monitoring of pregnancy.

In the initial visit, the type of physical activity will be evaluated by filling in the international physical activity questionnaire (IPAQ).

ELIGIBILITY:
Inclusion Criteria:

* To go to the Maternal Education program.
* Give your written consent to participate in the study.
* Singleton pregnancy.
* Low-risk pregnancy.
* No contraindication to physical exercise.
* Age equals or more than 18 years old.

Excusion Criteria:

* Pregnant women with poor pregnancy control.
* Difficulty in speaking or understanding Spanish.
* Required a C-section during delivery.
* Refusal to participate in the study.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-12-27 (Actual)

PRIMARY OUTCOMES:
Changes in the presence of pelvic floor injuries during childbirth after a Pilates Method program | Between the eighth and tenth day after birth
  Decrease in the number of episiotomies and perineal tears

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Feria-Ramírez, CNM, Principal Investigator — University of Huelva
Locations (1):
- Carmen Feria Ramírez, Lepe, Huelva, Spain

IPD SHARING:
Plan to Share IPD: Yes
The individual data will be available after deidenttification (text, tables, figures and appendices) to those researchers who provide a methodologically sound proposal and for meta-analysis.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available after the end of the study until one year the article publication.
Access Criteria: To obtain the data, a proposal must be sent to Carmen.feria@denf.uhu.es. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Almagiá E. Influencia del estado emocional en la salud física. Terapia psicológica. 2003; 21(1): 38.
- [Background] Aguiar M, Farley A, Hope L, Amin A, Shah P, Manaseki-Holland S. Birth-Related Perineal Trauma in Low- and Middle-Income Countries: A Systematic Review and Meta-analysis. Matern Child Health J. 2019 Aug;23(8):1048-1070. doi: 10.1007/s10995-019-02732-5. PMID 30915627
- [Background] Dieb AS, Shoab AY, Nabil H, Gabr A, Abdallah AA, Shaban MM, Attia AH. Perineal massage and training reduce perineal trauma in pregnant women older than 35 years: a randomized controlled trial. Int Urogynecol J. 2020 Mar;31(3):613-619. doi: 10.1007/s00192-019-03937-6. Epub 2019 Apr 2. PMID 30941442
- [Background] Graham ID, Carroli G, Davies C, Medves JM. Episiotomy rates around the world: an update. Birth. 2005 Sep;32(3):219-23. doi: 10.1111/j.0730-7659.2005.00373.x. PMID 16128977
- [Background] Jansson MH, Nilsson K, Franzen K. Development and validation of a protocol for documentation of obstetric perineal lacerations. Int Urogynecol J. 2019 Dec;30(12):2069-2076. doi: 10.1007/s00192-019-03915-y. Epub 2019 Mar 19. PMID 30888454
- [Background] Jiang H, Qian X, Carroli G, Garner P. Selective versus routine use of episiotomy for vaginal birth. Cochrane Database Syst Rev. 2017 Feb 8;2(2):CD000081. doi: 10.1002/14651858.CD000081.pub3. PMID 28176333
- [Background] Latorre GFS, de Fraga R, Seleme MR, Mueller CV, Berghmans B. An ideal e-health system for pelvic floor muscle training adherence: Systematic review. Neurourol Urodyn. 2019 Jan;38(1):63-80. doi: 10.1002/nau.23835. Epub 2018 Oct 30. PMID 30375056
- [Background] Mączka M, Sass A. Pilates and mobilization methods in therapy for low back pain among pregnant women. Journal of Exercise Science & Fitness. 2017; 7(8): 473-488.
- [Background] Boix-Vilella S, León-Zarceño E, Serrano-Rosa MA. Evidencias de la práctica Pilates sobre la salud mental de personas sanas. Rev Universidad y Salud. 2017; 19(2): 301-308.
- [Background] Bozkurt M, Yumru AE, Sahin L. Pelvic floor dysfunction, and effects of pregnancy and mode of delivery on pelvic floor. Taiwan J Obstet Gynecol. 2014 Dec;53(4):452-8. doi: 10.1016/j.tjog.2014.08.001. PMID 25510682
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Cruz-Ferreira A, Fernandes J, Laranjo L, Bernardo LM, Silva A. A systematic review of the effects of pilates method of exercise in healthy people. Arch Phys Med Rehabil. 2011 Dec;92(12):2071-81. doi: 10.1016/j.apmr.2011.06.018. Epub 2011 Oct 24. PMID 22030232
- [Background] Culligan PJ, Scherer J, Dyer K, Priestley JL, Guingon-White G, Delvecchio D, Vangeli M. A randomized clinical trial comparing pelvic floor muscle training to a Pilates exercise program for improving pelvic muscle strength. Int Urogynecol J. 2010 Apr;21(4):401-8. doi: 10.1007/s00192-009-1046-z. Epub 2010 Jan 22. PMID 20094704
- [Background] Davidson K, Jacoby S, Brown MS. Prenatal perineal massage: preventing lacerations during delivery. J Obstet Gynecol Neonatal Nurs. 2000 Sep-Oct;29(5):474-9. doi: 10.1111/j.1552-6909.2000.tb02768.x. PMID 11012126
- [Background] Dias NT, Ferreira LR, Fernandes MG, Resende APM, Pereira-Baldon VS. A Pilates exercise program with pelvic floor muscle contraction: Is it effective for pregnant women? A randomized controlled trial. Neurourol Urodyn. 2018 Jan;37(1):379-384. doi: 10.1002/nau.23308. Epub 2017 May 23. PMID 28543751
- [Background] D'Souza JC, Monga A, Tincello DG. Risk factors for perineal trauma in the primiparous population during non-operative vaginal delivery. Int Urogynecol J. 2020 Mar;31(3):621-625. doi: 10.1007/s00192-019-03944-7. Epub 2019 May 2. PMID 31049642
- [Background] Escuriet R, Pueyo MJ, Perez-Botella M, Espada X, Salgado I, Gomez A, Biescas H, Espiga I, White J, Fernandez R, Fuste J, Ortun V. Cross-sectional study comparing public and private hospitals in Catalonia: is the practice of routine episiotomy changing? BMC Health Serv Res. 2015 Mar 11;15:95. doi: 10.1186/s12913-015-0753-z. PMID 25889079
- [Background] Guzmán P, Díaz AM, Gómez D, Guzmán R, Guzmán A. Actuación del fisioterapeuta en el tratamiento integral de la embarazada. Nure Investigación. 2013; 2(63): 1-8.
- [Background] Howard D, Makhlouf M. Can pelvic floor dysfunction after vaginal birth be prevented? Int Urogynecol J. 2016 Dec;27(12):1811-1815. doi: 10.1007/s00192-016-3117-2. Epub 2016 Aug 15. PMID 27525694
- [Background] Hyakutake MT, Han V, Cundiff GW, Baerg L, Koenig NA, Lee T, Geoffrion R. Pelvic Floor Health Education: Can a Workshop Enhance Patient Counseling During Pregnancy? Female Pelvic Med Reconstr Surg. 2016 Sep-Oct;22(5):336-9. doi: 10.1097/SPV.0000000000000285. PMID 27171319
- [Background] Kyvernitakis I, Kohler C, Schmidt S, Misselwitz B, Grossmann J, Hadji P, Kalder M. Impact of maternal body mass index on the cesarean delivery rate in Germany from 1990 to 2012. J Perinat Med. 2015 Jul;43(4):449-54. doi: 10.1515/jpm-2014-0126. PMID 24914711
- [Background] Leon-Larios F, Corrales-Gutierrez I, Casado-Mejia R, Suarez-Serrano C. Influence of a pelvic floor training programme to prevent perineal trauma: A quasi-randomised controlled trial. Midwifery. 2017 Jul;50:72-77. doi: 10.1016/j.midw.2017.03.015. Epub 2017 Mar 27. PMID 28391147
- [Background] Llewellyn H, Konstantaki M, Johnson MI, Francis P. The Effect of a Pilates Exercise Programme on Perceived Functional Disability and Pain Associated with Non-Specific Chronic Low Back Pain. MOJ Yoga & Physical Therapy. 2017; 2(1): 00013.
- [Background] López M, Palacio M, del Pino M, Puig M, Bataller E, Espuña M. Protocolo: lesiones perineales de origen obstétrico. Diagnóstico, tratamiento y seguimiento. Servei de Medicina Maternofetal. Barcelona. Institut Clínic de Ginecologia, Obstetrícia i Neonatologia, Hospital Clínic de Barcelona. 2014.
- [Background] Navarro CL, Luján MI. Nuevos sistemas de comunicación del método Pilates en embarazo y puerperio. Revista Española de Comunicación en Salud. 2017; 8(1): 20-28.
- [Background] Neels H, Wyndaele JJ, Tjalma WA, De Wachter S, Wyndaele M, Vermandel A. Knowledge of the pelvic floor in nulliparous women. J Phys Ther Sci. 2016 May;28(5):1524-33. doi: 10.1589/jpts.28.1524. Epub 2016 May 31. PMID 27313364
- [Background] Oblasser C, McCourt C, Hanzal E, Christie J. Vibrating vaginal balls to improve pelvic floor muscle performance in women after childbirth: a protocol for a randomised controlled feasibility trial. J Adv Nurs. 2016 Apr;72(4):900-14. doi: 10.1111/jan.12868. Epub 2015 Dec 28. PMID 26708615
- [Background] Oktaviani I. Pilates workouts can reduce pain in pregnant women. Complement Ther Clin Pract. 2018 May;31:349-351. doi: 10.1016/j.ctcp.2017.11.007. Epub 2017 Nov 16. PMID 29173892
- [Background] Organización Mundial de la Salud.Cuidados en el parto normal: una guía práctica. Revista Hospital Materno Infantil Ramón Sardá. 1999; 18: 78-80.
- [Background] Pierce H, Perry L, Gallagher R, Chiarelli P. Pelvic floor health: a concept analysis. J Adv Nurs. 2015 May;71(5):991-1004. doi: 10.1111/jan.12628. Epub 2015 Feb 10. PMID 25675895
- [Background] Rodriguez-Diaz L, Ruiz-Frutos C, Vazquez-Lara JM, Ramirez-Rodrigo J, Villaverde-Gutierrez C, Torres-Luque G. Effectiveness of a physical activity programme based on the Pilates method in pregnancy and labour. Enferm Clin. 2017 Sep-Oct;27(5):271-277. doi: 10.1016/j.enfcli.2017.05.008. Epub 2017 Jul 6. English, Spanish. PMID 28689647
- [Background] Sarpkaya D.S., Yalvaç M. & Vural G. The effect of pregnancy Pilates-assisted childbirth preparation training on childbirth fear and neonatal outcomes: a quasi-experimental/quantitative research. Quality & Quantitive. 2018; 1-13.
- [Background] Shaban MM, Bassiouny YA, Elzahaby IM, Hassan AA. Body mass index and labour outcome in Egyptian women. J Obstet Gynaecol. 2014 Apr;34(3):248-50. doi: 10.3109/01443615.2013.844113. Epub 2013 Dec 2. PMID 24294988
- [Background] Smith LA, Price N, Simonite V, Burns EE. Incidence of and risk factors for perineal trauma: a prospective observational study. BMC Pregnancy Childbirth. 2013 Mar 7;13:59. doi: 10.1186/1471-2393-13-59. PMID 23497085
- [Background] Wells C, Kolt GS, Bialocerkowski A. Defining Pilates exercise: a systematic review. Complement Ther Med. 2012 Aug;20(4):253-62. doi: 10.1016/j.ctim.2012.02.005. Epub 2012 Mar 13. PMID 22579438
- [Background] Zimmo K, Laine K, Vikanes A, Fosse E, Zimmo M, Ali H, Thakar R, Sultan AH, Hassan S. Diagnosis and repair of perineal injuries: knowledge before and after expert training-a multicentre observational study among Palestinian physicians and midwives. BMJ Open. 2017 Apr 7;7(4):e014183. doi: 10.1136/bmjopen-2016-014183. PMID 28389490
- [Background] Rise E, Bo K, Nystad W. Is there any association between abdominal strength training before and during pregnancy and delivery outcome? The Norwegian Mother and Child Cohort Study. Braz J Phys Ther. 2019 Mar-Apr;23(2):108-115. doi: 10.1016/j.bjpt.2018.06.006. Epub 2018 Jul 6. PMID 30017257
- [Background] Uccella S, Manzoni P, Marconi N, Toscani C, Biasoli S, Cianci S, Franchi M, Sorice P, Bertoli F, Zorzato PC, Gallina D, Ghezzi F, Serati M. Impact of Sport Activity and Physical Exercise on Obstetrical and Perineal Outcomes at Delivery: A Prospective Study. Am J Perinatol. 2019 Jul;36(S 02):S83-S90. doi: 10.1055/s-0039-1691816. Epub 2019 Jun 25. PMID 31238366
- [Background] Verghese TS, Champaneria R, Kapoor DS, Latthe PM. Obstetric anal sphincter injuries after episiotomy: systematic review and meta-analysis. Int Urogynecol J. 2016 Oct;27(10):1459-67. doi: 10.1007/s00192-016-2956-1. Epub 2016 Feb 19. PMID 26894605
- [Background] Waddington H, Aloe AM, Becker BJ, Djimeu EW, Hombrados JG, Tugwell P, Wells G, Reeves B. Quasi-experimental study designs series-paper 6: risk of bias assessment. J Clin Epidemiol. 2017 Sep;89:43-52. doi: 10.1016/j.jclinepi.2017.02.015. Epub 2017 Mar 27. PMID 28351693
- [Derived] Feria-Ramirez C, Gonzalez-Sanz JD, Molina-Luque R, Molina-Recio G. The Effects of the Pilates Method on Pelvic Floor Injuries during Pregnancy and Childbirth: A Quasi-Experimental Study. Int J Environ Res Public Health. 2021 Jun 30;18(13):6995. doi: 10.3390/ijerph18136995. PMID 34208859
- See also: Proceso Asistencia Integrado embarazo, parto y puerperio — https://www.juntadeandalucia.es/export/drupaljda/salud_5af1956fa966b_embarazo_parto_puerperio_septiembre_2014.pdf

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-10): https://cdn.clinicaltrials.gov/large-docs/02/NCT04431102/Prot_SAP_000.pdf
  • Informed Consent Form (2018-10-10): https://cdn.clinicaltrials.gov/large-docs/02/NCT04431102/ICF_001.pdf